CLINICAL TRIAL: NCT04757259
Title: An Expanded Access Protocol for Patients Who Completed Study 13-601 and Continue to Clinically Benefit From Cerdulatinib
Brief Title: Expanded Access Program for Participants Who Completed Study 13-601 and Continue to Clinically Benefit From Cerdulatinib
Status: No longer available | Type: Expanded Access
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-605
Record Dates: First submitted 2021-02-10; First posted 2021-02-17 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Relapsed/Refractory Chronic Lymphocytic Leukemia; Non-hodgkin's Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — 4-(cyclopropylamino)-2-((4-(4-(ethylsulfonyl)piperazin-1-yl)phenyl)amino)pyrimidine-5-carboxamide

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: cerdulatinib — Participants will receive oral cerdulatinib at the starting dose he or she was receiving at completion of Study 13-601 (30, 25, 20, or 15 milligrams [mg] twice daily [BID]).
  Other Names: PRT062070

SUMMARY:
This expanded access program will provide continued access to cerdulatinib to eligible participants who experienced clinical benefit from cerdulatinib in Study 13-601 (NCT01994382) and who otherwise meet the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed Portola Study 13-601 and wishes to continue treatment with cerdulatinib.
* In the opinion of the Investigator, the potential benefit to the participant of continuing to receive cerdulatinib outweighs the risks.
* Female participants of childbearing potential and male participants must agree to continue to abstain from sexual intercourse or to remain on an effective method of contraception during treatment and for 90 days following the last dose of protocol therapy (examples of effective methods of contraception include oral contraceptives or double barrier methods, such as condom plus spermicide or condom plus diaphragm).
* Participant must be willing to give written informed consent and be able to adhere to dose and visit schedules.

Exclusion Criteria:

* Participant requires chronic treatment with a strong CYP3A4 inhibitor or inducer.
* Participant has a known hypersensitivity to any of the components of cerdulatinib.
* Participant is female and is breast-feeding, pregnant, or intends to become pregnant.
* Participant is participating in any therapeutic clinical study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult